CLINICAL TRIAL: NCT02749942
Title: The RISCAID Study: Remote ISchemic Conditioning for Angiopathy In Diabetes
Brief Title: RISCAID Study: Remote ISchemic Conditioning for Angiopathy In Diabetes
Acronym: RISCAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); German Diabetes Center (Other)
Responsible Party: Principal Investigator, Peter Rossing, Professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RISCAID
Record Dates: First submitted 2016-04-04; First posted 2016-04-25 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Diabetes; Remote Ischemic Conditioning; Neuropathy; Angiopathy
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AutoRIC: Remote Ischemic Conditioning (Active Comparator): Daily cuff treatment of arm with 4 cycles of 5 minute forearm ischemia/reperfusion (200 mmHG of pressure) on top of standard care.
  Interventions: Device: AutoRIC: Remote Ischemic Conditioning
- AutoRIC: Sham device treatment (Sham Comparator): Daily sham device treatment of arm, 4 cycles of 5 minute (0 mmHG of pressure) on top of standard care. No ischemia induced.
  Interventions: Device: AutoRIC: Sham device treatment

INTERVENTIONS:
Device: AutoRIC: Remote Ischemic Conditioning — 4 cycles of 5 minute forearm ischemia/reperfusion (200 mmHG) using the reusable fully automated RIC device "AutoRIC" from CellAegis Devices, Canada
  Arms: AutoRIC: Remote Ischemic Conditioning
Device: AutoRIC: Sham device treatment — 4 cycles of 5 minute forearm sham treatment (no ischemia/reperfusion, 0 mmHG pressure) with the reusable fully automated RIC device "AutoRIC" from CellAegis Devices, Canada
  Arms: AutoRIC: Sham device treatment

SUMMARY:
Objective The objective of this study is to investigate if long-term ambulatory remote ischemic conditioning can improve symptoms and signs of peripheral arterial disease in patients with type 2 diabetes.

Background Peripheral arterial disease (PAD) is a vast socioeconomic challenge in the community of diabetes patients, causing foot ulcers and lower extremity amputations. The main treatment option for the complication is operative revascularisation. Thus there is a need for new treatment modalities for diabetes patients with PAD.

Remote ischemic conditioning (RIC) is at non-invasive non-pharmacological treatment which has been shown to attenuate tissue damage caused by ischemia e.g. in hearts subjected to ischemia. RIC treatment consists of brief repetitive periods of ischemia induced in an extremity e.g. an arm. Recent findings show that six week RIC treatment improves healing of diabetic foot ulcers, suggesting a possible effect on the underlying pathological causes of ulcers e.g. PAD.

Hypothesis The investigators hypothesize that RIC treatment can improve markers of inflammation, vascular and neuronal function and the sense of empowerment in type 2 diabetes patients with reduced peripheral blood supply.

Aim to conduct a single center double-blinded randomized placebo controlled study investigating the efficacy of home based 12-week RIC treatment on markers of vascular, neuronal function, inflammation and serum lipid composition in 40 type 2 diabetes patients from Steno Diabetes Center with non-critical PAD.

to qualitatively investigate the experience of empowerment related to the use of Remote Ischemic Conditioning (RIC) treatment and the mechanisms affecting if and how participants take up the RIC treatment.

DETAILED DESCRIPTION:
Objective The driving objective of this study is to investigate if long-term ambulatory remote ischemic conditioning can improve symptoms and signs of peripheral arterial disease and the sense of empowerment in patients with type 2 diabetes.

Background Peripheral arterial disease (PAD) is vast challenge in the community of diabetes patients. The prevalence of PAD in diabetes patients exceeds that of non-diabetic individuals and is estimated to be about 26% in diabetes patients over 65 years of age and 71% in patients over 70 years . PAD is the major cause of foot ulcers and lower extremity amputations, which has great socioeconomic implications . The main treatment option for the complication is operative revascularisation which in diabetes patient is associated with increased rates of complication and mortality compared to non-diabetes patients . Pharmacological treatment with e.g. anti-platelet drugs in patients with PAD has shown effect on walking distance has not been indorsed as standard treatment.

Thus there is a need for new treatment options for diabetes patients with PAD. Remote ischemic conditioning (RIC) is a non-invasive non-pharmacological treatment that has been shown to attenuate tissue damage caused by ischemia, reducing infarct size in patients with acute myocardial infarction , reducing organ damage in patient undergoing transplantation and having neuroprotective effects in patients with stroke .

RIC treatment consists of brief repetitive periods of ischemia induced in an extremity e.g. an arm. It is believed that the effect of RIC is mediated through both neuronal and humoral pathways, however the mechanisms behind are not fully understood.

RIC has been shown to have beneficial effects by attenuating platelet activation and aggregation, improving endothelial function , improvement of microcirculation , down-regulation of neutrophil function , down-regulation of inflammatory gene expression , improving mitochondrial function and inducing changes in serum lipid composition One of few long-term RIC treatment studies has shown that twice daily RIC treatment for 300 days is feasible. The study showed that RIC could reduce the recurrence of stroke

. No studies are presently investigating the effect of long-term RIC on PAD in diabetes patients (Clinicaltrials.gov search 22nd of October 2015), the concept has however recently been presented in the literature . Two studies have addressed the acute effect of one RIC treatment on walking distance in non-diabetic patients with claudication. The results were inconclusive due to small sample sizes, but a trend towards improvement was shown. It is however likely that long-term RIC treatment is needed to show a beneficial effect of RIC on the pathology behind claudication - vascular and neuronal damage.

Hypothesis We hypothesize that the long-term RIC treatment can improve PAD. PAD is caused by both micro- and macrovascular deficits. Reduced microvascular circulation can lead to distal nerve damage which in turn can both reduce peripheral circulation and cause tissue degeneration. Reduced macro vascular function is a direct cause of peripheral ischemia (2). It is possible that RIC could attenuate the pathophysiological processes in the micro- and microvasculature related to PAD by the abovementioned mechanisms and thereby improving of both neuronal and vascular function.

Thus the present clinical evidence of the beneficial effects of RIC may be translated into a new safe and simple non-invasive non-pharmacological treatment of PAD in diabetes patients, preventing progression to critical ischemia and amputation.

We also hypothesize that home-based and self-administered RIC treatment can improve the sense of empowerment in patients with non-critical peripheral arterial disease and type 2 diabetes.

Aims and Methods

Primary aim:

to study the underlying mechanisms of the effects of long-term ambulatory RIC by investigating the effect on vascular function, neuronal function, markers of inflammation, oxidative stress and endothelial dysfunction and lipidomic profiles.

Secondary aim to study the the experience of the use of RIC treatment and with focus on barriers that affect the uptake of the RIC treatment, and the effects of treatment on life quality and empowerment.

Study design The study will consist of a single-center randomised double blinded placebo controlled trial.

The trial will be performed to investigate the beneficial effects of RIC treatment on the study outcomes described below. The RIC treatment duration will be 12 weeks and 40 patients from the Steno Diabetes Center will be included in the trial. All tests and analyses will performed at Steno Diabetes Center expect for markers of inflammation and oxidative stress which will be performed at Dept. of inflammation, German Diabetes Center and institute of Clinical Diabetology, German Diabetes Center. All necessary facilities are available at the study sites.

Most present knowledge of the beneficial effects of RIC listed above has come from short term trials (duration = 1 day. 20 days for one study) with small populations (n ≤ 40). Thus it is plausible that the study setup will yield significant differences in outcomes between the study arms. The study may also indicate if changes in outcomes will occur post RIC treatment.

For the qualitative part of the study relevant questionnaires will be filled out at baseline and end-of trial. In addition 15 random patients will be asked to attend "think-aloud" interviews within the last 4 weeks of treatment.

Power calculation RIC has shown to increase tissue oxygen tension (a measure of microcirculation) in a short-term study we hypothesize that RIC treatment will increase tissue oxygen tension in the feet (Primary outcome) by 13% (SD = 10%). With 90% power and a two sided significance level of 0.05 the sample size needed to detect this change is 16 in each group - 32 participants in total. Taking a drop-out ratio of 10% into account and given the inaccurate nature of this power calculation the sample size of the study will be 20 patients in each group.

Statistics The effects of treatment on outcome measures will be estimated by using complete-case logistic regression analyses. If needed outcome variables will be log-transformed using the natural logarithm to meet model assumptions of the distribution of the model residuals if necessary. Interactions between sex and all determinants will be investigated in all models to investigate possible sex interactions differences. A level of significance of 5% will be used.

Analyses will be performed using SAS version 9.3 (SAS Institute, Cary, NC). Discontinuation of single person participation in study or cancellation of whole study The doctor responsible for the study can at any time discontinue the study for any reason e.g. for safety concerns. The responsible doctor can discontinue the participation of any single participant if informed consent is withdrawn, the a participant wants to get pregnant or get pregnant, if a participant does not follow the study protocol. A participant can withdraw his or her participation without justification at any time and this will not influence the treatment at Steno Diabetes Center of the participant.

Data storage All procedures and facilities for data handling and storage will follow the rules and regulations of Datatilsynet. Permission from Datatilsynet for collecting and storing the data will be sought prior to the study start.

All data from will be stored at the Steno Diabetes Center, Niels Steensens Vej 4, in Gentofte, Denmark. No person sensitive data will be shared with collaborator outside of Steno Diabetes Center. Data on analyses done at the German Diabetes Institute will be handle only by use of the patients trail number.

All data gathered on paper during the clinical examination will be stored in a locked archive at Steno Diabetes Center.

Publication Data is owned by the Steno Diabetes Center A/S. Positive (significant), negative (non-significant) and inconclusive results will be published as soon as it is scientifically justifiable.

Significance and perspectives If the project shows an effect of RIC on PAD the next step will to test the treatment method in a larger trial where walking distance will be the primary outcome. Also it is possible that patients with foot ulcers and patients with critical peripheral ischemia could benefit from the treatment.

RIC treatment could prove to be an attractive non-pharmacological non-surgical treatment option for a large population of diabetes patients. The trial will result in 5 publications on the efficacy of RIC on neuronal function, on vascular function, on lipidomic profiles, on marker of inflammation and oxidative stress (Tentative titles of articles are listed in Appendix 3) and patient empowerment and quality of life. The study is recommended by an independent Professor of Cardiology (Appendix 4).

Possible limitations It is debated whether or not diabetes can attenuated the efficacy of RIC treatment. Data from randomised clinical trials are conflicting . As the patients in the present study population will have some degree of neuropathy this may attenuate the effect of RIC on our outcomes. However a recent study has showed an effect of RIC on diabetic foot ulcers contradicting the above-mentioned hypothesis, as all diabetes patients with foot ulcers have some degree of neuropathy .

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age 40-80
* Complaints of claudication or reduced walking distance compared to equals
* Toe pressure from 40 mmHG to 70 mmHg

Exclusion Criteria:

* Foot ulcer
* Peripheral gangrene or infection
* Toe pressure < 40 mmHg or > 90 mmHg
* Heart failure
* Pregnancy
* Treatment with anti-platelet drugs besides acetylsalicylic acid
* Cancer
* Chronic obstructive pulmonary disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Peripheral tissue oxygen oxygenation of dorsal part of foot | Change from baseline to 12 weeks of treatment
  Transcutaneous oxygen tension

SECONDARY OUTCOMES:
Toe Pressure | At baseline and fter 12 weeks of treatment and 4 weeks post treatment
  pressure
Central vasculopathy | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Arterial stiffness assessed and central blood pressure by pulse wave velocity measures
Glycocalyx assessment | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Arterial function assessed by sublingual capillary density and perfused boundary region
Cardiovascular autonomic neuropathy, E/I ratio | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Cardiovascular reflex test: E/I ratio
Peripheral autonomic function | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Peripheral small-fibre sympathetic function by sudomotor function testing assessed by electrochemical skin conductance
Peripheral nerve conduction function | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Sural nerve conduction velocity
Sensory peripheral neuropathy, vibration | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  toe vibration sensation threshold
Sensory peripheral neuropathy, light touch | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  light touch assessed by 10 gram monofilament
Sensory peripheral neuropathy, pain sensation | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  pain sensation assessed by pin prick
symptoms of neuropathy | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Minnesota Neuropathy Screening Instrument questionnaire
Cardiovascular autonomic neuropathy; 30/15 ratio | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Cardiovascular autonomic reflex test; E/I ratio
Cardiovascular autonomic neuropathy, Valsalva maneuvre | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Cardiovascular autonomic reflex test; Valsalva maneuvre
Cardiovascular Autonomic neuropathy; Heart rate variability | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  5 minute resting hear rate variability measure.

OTHER OUTCOMES:
Serum markers of inflammation, 1 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  hsCRP
Serum markers of vascular function, 1 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  thiobarbituric acid reactive substances (TBARS)
Serum markers of kidney function | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  eGFR
Cardiometabolic markers, 1 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Cholesterol profile
Metabolomic markers | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Spectrometry-based profiling of the serum lipidome
Assessment of quality of life and empowerment, 1 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Diabetes Empowerment Scale (DES)
Serum markers of inflammation, 2 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  interleukin-6
Serum markers of inflammation, 3 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  interleukin-1beta
Serum markers of inflammation, 4 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  interleukin-1RA
Serum markers of inflammation, 5 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  adiponectin
Serum markers of vascular function, 2 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  thiobarbituric acid reactive substances (TBARS)
Serum markers of vascular function, 3 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  extracellular superoxide dismutase-3 (SOD3)
Serum markers of vascular function, 4 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  glutathione (GSH) soluble vascular cell adhesion molecule-1 (sVCAM-1)
Serum markers of vascular function, 5 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  soluble intercellular adhesion molecule-1 (sICAM-1)
Serum markers of vascular function, 6 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  endothelial nitric oxide synthase
Serum markers of vascular function, 7 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  cyclooxygenase
Serum markers of vascular function, 8 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  prostacyclin synthase
Serum markers of vascular function, 9 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  thromboxane synthase
Serum markers of vascular function, 10 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  endothelin receptor A/B
Serum markers of vascular function, 11 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  plasma NO metabolites nitrite and nitrate
Serum markers of vascular function, 12 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  prostacyclin
Serum markers of vascular function, 13 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  thromboxane
Serum markers of vascular function, 14 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  endothelin-1
Marker of kidney function | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Urine albumin creatinine ratio.
Cardiometabolic markers, 2 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Serum Triglycerides
Cardiometabolic markers, 3 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Serum HbA1C
Assessment of quality of life and empowerment, 2 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Who-Five Well-being Index
Assessment of quality of life and empowerment, 3 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  Diabetes Distress Scale
Assessment of quality of life and empowerment, 4 | At baseline and 1, 4 and 12 weeks of treatment and 4 weeks post treatment
  WHO-5

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Professor, Principal Investigator — Head of department
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No
To ensure data security no data will be shared outside the study group

REFERENCES:
- [Derived] Hansen CS, Jorgensen ME, Fleischer J, Botker HE, Rossing P. Efficacy of Long-Term Remote Ischemic Conditioning on Vascular and Neuronal Function in Type 2 Diabetes Patients With Peripheral Arterial Disease. J Am Heart Assoc. 2019 Jul 2;8(13):e011779. doi: 10.1161/JAHA.118.011779. Epub 2019 Jun 19. PMID 31215299